CLINICAL TRIAL: NCT02637050
Title: EMEA CTEPH Registry: An International Prospective Registry Investigating the Epidemiology, Diagnosis and Treatment of CTEPH Patients in EMEA Countries
Brief Title: A Study Investigating Routine Practice of Chronic Thromboembolic Pulmonary Hypertension Management in EMEA Countries
Acronym: EMEA CTEPH
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 18303; AD 1502 (Other: Company Internal)
Record Dates: First submitted 2015-12-04; First posted 2015-12-22 (Estimated); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Hypertension, Pulmonary
Keywords: Type IV Pulmonary Hypertension; Chronic Thromboembolic Pulmonary Hypertension; CTEPH
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CTEPH Patients: Patients with confirmed diagnosis of CTEPH
  Interventions: Other: Standard of care

INTERVENTIONS:
Other: Standard of care — At the discretion of the attending physician.

SUMMARY:
The aim of the registry is the assessment of the diagnosis and treatment of CTEPH (Chronic Thromboembolic Pulmonary Hypertension) in EMEA (Europe/Middle East/Africa) countries.

ELIGIBILITY:
Inclusion Criteria:

* Female and male patients ≥ 18 years of age, diagnosed with CTEPH regardless of the current treatment
* Availability of a signed informed consent
* WHO Pulmonary Hypertension clinical classification Group IV (CTEPH):

  1. Right heart catheterization (RHC) results that are in line with both of the following haemodynamic levels:

     * Mean pulmonary arterial pressure (PAP) ≥ 25 mmHg at rest
     * Pulmonary arterial wedge pressure (PAWP) ≤ 15 mmHg
  2. Confirmation of CTEPH diagnosis by one of the following as recommended by standard guidelines:

     * At least 1 (segmental) perfusion defect(s) in ventilation/perfusion (V/Q) scan or
     * Pulmonary artery obstruction seen by MDCT (multidetector computed tomography) angiography or
     * Pulmonary artery obstruction seen by conventional pulmonary cineangiography (In case of suspicion/diagnosis of 'sub-acute' Pulmonary Embolism: Patients who are treated with anti-coagulation for at least 3 months before diagnosis of CTEPH)

Exclusion Criteria:

* Patients with an underlying medical disorder with an anticipated life expectancy less than 6 months
* Any medical condition which, in the opinion of the investigator, could jeopardize the safety of the patient or his/her compliance in the study, or otherwise make the patient inappropriate for study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CTEPH (Chronic Thromboembolic Pulmonary Hypertension) patients in Expert PH (Pulmonary Hypertension) centers
Sampling Method: Non-Probability Sample
Enrollment: 231 (Actual)
Dates: Start 2016-03-03 (Actual); Primary Completion 2020-07-03 (Actual); Study Completion 2020-09-17 (Actual)

PRIMARY OUTCOMES:
The clinical functional parameters of CTEPH patients will be assessed by evaluating the change in measures of 6MWD between initial and final visit | Up to 3 years
  6MWD (6 Minutes Walking Distance)
The clinical functional parameters of CTEPH patients will be assessed by evaluating the change in measures of WHO Functional Class between initial and final visit | Up to 3 years
  WHO Functional class (World Health Organization Functional Class)
The haemodynamics parameters of CTEPH patients will be assessed by evaluating the change in measures of PVR between initial and final visit | Up to 3 years
  PVR (Pulmonary Vascular Resistance)
The haemodynamics parameters of CTEPH patients will be assessed by evaluating the change in measures of Cardiac Index (CI) between initial and final visit | Up to 3 years
  CI (Cardiac Index)
The haemodynamics parameters of CTEPH patients will be assessed by evaluating the change in measures of mPAP between initial and final visit | Up to 3 years
  mPAP (mean Pulmonary Arterial Pressure)

SECONDARY OUTCOMES:
Eligibility for PEA | Up to 3 years
  At inclusion, information will be collected for each patient regarding their eligibility for PEA. If eligible, details about the PEA will be recorded; if not eligible, further information will be collected to understand why the patient was not eligible.
Rate of recurrent to persistent subtypes after Pulmonary Endarterectomy | Up to 3 years
  Not yet assessable/Recurrent/Residual
Time span between onset of symptoms and CTEPH diagnosis | Up to 3 years
Usage of diagnostic tools of CTEPH patients (Y/N) | Up to 3 years
Rate of Pulmonary Hypertension treatments prior to CTEPH diagnosis, at the time of CTEPH diagnosis and at the time of first visit | Up to 3 years
Treatment duration with Pulmonary Hypertension treatments prior to CTEPH diagnosis, at the time of CTEPH diagnosis and at the time of first visit | Up to 3 years
Changes in CTEPH treatment during the study period | Up to 3 years
Number of patients eligible for Pulmonary endarterectomy | Up to 3 years
NT-proBNP (N-terminal Propeptide Brain Natriuretic Peptide) levels | Up to 3 years
Mortality due to CTEPH and CTEPH related complications | Up to 3 years
Number of healthcare professional visits due to CTEPH and CTEPH related complications | Up to 3 years
The total number of days of hospitalization due to CTEPH and CTEPH related complications | Up to 3 years
Number of patients eligible for Balloon Pulmonary Angioplasty | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (6):
- Multiple Locations, Kazakhstan
- Multiple Locations, Kyrgyzstan
- Multiple Locations, Lebanon
- Multiple Locations, Russia
- Multiple Locations, Saudi Arabia
- Multiple Locations, Turkey (Türkiye)

REFERENCES:
- [Derived] Ongen HG, Akdeniz B, Duzenli MA, Chernyavsky A, Dabar G, Idrees M, Khludeeva E, Kultursay H, Lukianchikova V, Martynyuk T, Mogulkoc N, Mukarov MA, Mutlu B, Okumus G, Omarov A, Onen ZP, Sakkijha H, Shostak N, Simakova M, Tokgozoglu L, Tomskaya T, Yildirim H, Zateyshchikov D, Hechenbichler K, Kessner S, Schauerte I, Turgut N, Vogtlander K, Aldalaan A; CTEPH EMEA Registry Investigators. Diagnosis and Treatment Patterns of Chronic Thromboembolic Pulmonary Hypertension in Russia, Kazakhstan, Turkey, Lebanon, and Saudi Arabia: A Registry Study. Drugs Real World Outcomes. 2024 Mar;11(1):149-165. doi: 10.1007/s40801-023-00407-w. Epub 2024 Feb 21. PMID 38381283